CLINICAL TRIAL: NCT06379698
Title: Effects of a Personalized or Generic Three-dimensional Tumoral Kidney Model on Patient Experience and Professional-patient Interactions, Before and After Partial Nephrectomy
Brief Title: Rein 3D PRINT PERSONALIZE
Acronym: R3DP-P
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2023/78
Record Dates: First submitted 2024-03-19; First posted 2024-04-23 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-04

CONDITIONS: Tumoral Kidney
Keywords: Renal-Cell Carcinoma; Nephron-Sparing Surgery; 3D Model; 3D Printing; Personalized Medicine; Literacy Questionnaire
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- personalized 3D kidney model (Active Comparator): exchange time with the personalized 3D model of the kidney to be operated on as information support
  Interventions: Other: personalized 3D model pré-opérative education
- generic 3D kidney model (Active Comparator): exchange time with the generic 3D model of the kidney to be operated on as information support
  Interventions: Other: generic 3D model pré-opérative education

INTERVENTIONS:
Other: personalized 3D model pré-opérative education — Before surgery, during a preoperative therapeutic education consultation, a personalized 3D models will be presented to the patients according to the allocated study group
  Arms: personalized 3D kidney model
Other: generic 3D model pré-opérative education — Before surgery, during a preoperative therapeutic education consultation, a generic 3D models will be presented to the patients according to the allocated study group
  Arms: generic 3D kidney model

SUMMARY:
The goal of this clinical trial is to compare preoperative information and patient experience using a personalized versus a generic 3D printed models of patients' tumoral kidney before and after nephron-sparing surgery. The main outcome measure will be based on semi-structured interviews with the patient and the carers.

DETAILED DESCRIPTION:
The use of tools to decrease anxiety and enhance understanding prior to surgery is a key point in comprehensive care that is way not enough promoted for now.

A pilot study from 2015 demonstrated the benefits of using personalized 3D-printed kidney models as educational mediation tools during the pre-operative consultation of patients scheduled for robot-assisted partial nephrectomy. The patient's understanding of his pathology and of the surgery was thus facilitated, leading to greater satisfaction during treatment.

For personalized medicine, it is important to consider the heterogeneity in culture and social backgrounds of patients in the doctor-patient relationship. Measuring health literacy help to identify and describe this heterogeneity in patient profiles. Patients with low literacy levels have higher levels of anxiety, particularly regarding surgery, and poorer post-operative recovery. Some studies highlight the importance of improving patient understanding with strategies to improve patients' health literacy and information provided by carers.

The goal of this study is therefore to investigate the benefits of using a personalized 3D-printed kidney model versus a generic 3D-printed kidney model as a mediation tool, all along the care pathway, on patients' experience and their interactions with carers, before and after partial nephrectomy.

To achieve this aim, 60 patients planned for robot-assisted laparoscopic partial nephrectomy will be randomized, in a 1:1 ratio, between the use of a personalized 3D kidney model and a generic 3D kidney model.

3D models will be presented to the patients according to the allocated study group during a preoperative education consultation. All patients will complete questionnaires about their health literacy level, their knowledge of kidney anatomy and tumor and their satisfaction about the using 3D-printed kidney models as educational mediation tools. Semi-structured interviews will be conducted at three different times: between the first consultation with the surgeon and the preoperative education consultation, between this second consultation and the surgery and after the post-operative consultation.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Adult patients (≥ 18 years of age)
* Scheduled for surgical management by laparoscopic robotic-assisted partial nephrectomy (1st management for a unilateral or bilateral kidney tumor)
* Expressed consent for integration in the UroCCR database
* Expressed consent for participation in the Rein-3D Personalize study
* Patients affiliated or benefiting from social security system

Professionals:

* Professionals working with patients treated in the Urology, Andrology and Renal Transplant - Department of the Bordeaux University Hospital for at least two months prior to the implementation of 3D models
* Free, informed and signed consent

Exclusion Criteria:

Patients

* Metastatic at inclusion
* Previous renal cancer(s)
* Single kidney at time of inclusion
* No preoperative CT scan, or poor-quality CT scan unable to provide reliable 3D modeling
* Person under legal protection (safeguard of justice, guardianship or curatorship)
* Difficulty understanding and expressing oneself in French

Professionals

* Professionals on internship lasting less than 6 months
* Professionals with no contact with patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Qualitative assessment of patient experience 1 | between baseline and Day15 post-op
  Patient experience will be measured by a set of element including observations and 3 questionnaires described in outcome 1, outcome 2, outcome 3.
  Measurement of the progression in mean health literacy questionnaire score HLSEU-Q16 this questionnaire is a short version version of the European Health Literacy Survey Questionnaire (Sørensen et al., 2013), based on a model including 4 health information processing skills: accessing, understanding, evaluating and applying application of health information. The Items are scored from 'Strongly Disagree' to 'Strongly Agree', and from 'Cannot Do' to 'Very Easy'. The total score is produced by summing all items
Qualitative assessment of patient experience 2 | between baseline and Day15 post-op
  Patient experience will be measured by a set of element including observations and 3 questionnaires described in outcome 1, outcome 2, outcome 3.
  Measurement of the level of understanding of renal anatomy and surgical issues using the Bernhard et al. questionnaire.
  The knowledge questionnaire ( Bernhard 2016) consists of 4 parts: basic kidney physiology, basic kidney anatomy, tumor characteristics and planned surgical procedure. The patient answers 'False' , 'True' or 'Don't know'. The scores are calculated in each part by calculating the numbers of correct answers .
  These dimensions will be studied before and after the presentation of the model, and compared according to the model used.;
Qualitative assessment of patient experience 3 | between baseline and Day15 post-op
  Patient experience will be measured by a set of element including observations and 3 questionnaires described in outcome 1, outcome 2, outcome 3.
  Patient satisfaction is measured using the satisfaction questionnaire adapted from the Bernhard 2016 study. This measures how well the three-dimensional printed kidney model helped patients in learning " basic notions " about the kidney, and improving their understanding of : the disease, the scheduled surgery and the risk of complications related to the surgery. Each of the four dimensions is rated by a 10-point score ranging from 1 "no help at all" to 10 "great help". The average of the scores per dimension and an overall satisfaction score will be calculated and compared between the groups.

SECONDARY OUTCOMES:
Description of interactions between carers and patients | between baseline and Day15 post-op
  The description will be done according to the 3 D model used, specifying the aproach based on individual semi-directive interviews exploring patient experience, health education and health literacy as well as the vocabulary and content of the discourse employed.
Comparison of the evolution and frequency of terms used by patients in the 2 groups during their care. | between baseline and Day15 post-op
  The comparison will be done by evaluation of the evolution and frequency of terms used by patients : terms related to the pathology, the kidney model used, interactions with professionals in the care circuit
Studying the use of the 3D-printed kidney model introduced during the medical information consultation up to the post-operative visit by describing the life of the model throughout the entire care process | between baseline and Day 15 post-op
To study the level of understanding of renal anatomy and surgical issues according to the type of tool (personalized vs generic 3D printed model) | baseline ; between D-1 and Day-15 from surgery ; Day 15 post-op
  Level of understanding measured by the Bernhard et al questionnaire. This questionnaire consists of 4 parts: physiological and anatomical dimensions, knowledge of the disease and tumor characteristics, understanding of the surgical procedure and associated complication risks. These dimensions will be studied before and after the presentation of the model, and compared according to the model used. The final part of the questionnaire, based on an assessment of patient satisfaction, will be presented at the end of the post-operative consultation period
Comparison of the level of health literacy between the two groups at different times with changes in the average score on the literacy questionnaire (HLSEU-Q16: European Health Literacy Survey Questionnaire) | baseline ; Day-30 post-op
  This questionnaire is a short version version of the European Health Literacy Survey Questionnaire (Sørensen et al., 2013), based on a model including 4 health information processing skills: accessing, understanding, evaluating and applying application of health information . Patients respond on a 4 scale ranging from "very easy" to "very difficult". The overall score scales from 0 to 16 points. This score is used to determine 3 levels of literacy: unsatisfactory (0-8), average(9-12) and satisfactory (13-16).
Description of the changes perceived by carers in patients management in both group | between baseline and year 1 post baseline
  Qualitatively assessment of changes in practices following the integration of 3D models into the department's practices. This analysis will be based on interviews with professionals, describing their relationship with patients and their families.

CONTACTS AND LOCATIONS:
Overall Officials: Gaëlle MARGUE, Docteur, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pattou M, Masanet S, Jutand MA, Hoarau H, Sarrazin J, Pitout A, Richert L, Larribere H, Rubat Baleuri F, Jaffredo M, Ricard S, Faessel M, Sabatier J, Bernhard JC, Margue G. Effects of a personalized or generic three-dimensional tumoral kidney model on patient experience and caregiver-patient interactions, before and after partial nephrectomy, a randomized trial (Rein 3D Print Personalize-UroCCR 114). PLoS One. 2025 Aug 18;20(8):e0323515. doi: 10.1371/journal.pone.0323515. eCollection 2025. PMID 40824885